CLINICAL TRIAL: NCT03924583
Title: Diagnostic Reliability of Duplex Ultrasonography of the Venous System for Screening of Catheter-related Thrombosis Performed by a General Nurse
Brief Title: Duplex Ultrasonography Performed by Nurses
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Masaryk Hospital Krajská zdravotní a.s. (Other)
Responsible Party: Principal Investigator, Barbora Pakostová, M.D., Medical doctor, Masaryk Hospital Krajská zdravotní a.s.
Other Study IDs: 258/40
Record Dates: First submitted 2019-04-17; First posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Catheter Related Complication
MeSH Terms: interventions — Ultrasonography, Doppler, Duplex

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Duplex ultrasonography — Ultrasound examination of whole vena cava venous system with central venous catheter inserted, using duplex US method to detect catheter related thrombosis

SUMMARY:
Catheter-related thrombosis (CRT) has been found as the major complication of the established central venous catheter in intensive care unit (ICU) patients. Its reported incidence varies from 5 to 66 %. Although most cases are asymptomatic, in up to 10 - 15 % of the patients pulmonary embolism occurs. In addition, CRT is associated with the risk of infection, post-thrombotic syndrome and with general disruption of the management of the underlying disease. The most accessible diagnostic method for CRT recognition is duplex ultrasonography. However, screening of CRT by duplex ultrasonography is not common approach in ICUs. Normally, duplex ultrasonography is performed by physicians. In this setting, implementation of the screening in ICU would be time consuming and practically unrealizable. Delegating this competence to ICU nurses can increase availability of this screening method.

Therefore, as a first step, investigators decided to perform a validation clinical study to verify the diagnostic accuracy of duplex ultrasonography of the venous system for CRT screening performed by a general nurse.

DETAILED DESCRIPTION:
Approximately 150 patients with central venous catheter will be enrolled in this study.

Investigators:

1. General nurses - trained and able to perform duplex ultrasonography examination of venous circulation
2. Doctors - experienced specialists in intensive care or urgent medicine

Every patient with central venous catheter enrolled in clinical study is examined with duplex ultrasonography within 24 hours by both investigators, doctor and nurse. Each examination includes ultrasonography of a whole vena cava venous system with central venous catheter, bilaterally. Results of both examinations are blinded until the end of study, with one exception. In case of positive result - catheter related thrombosis is present, investigator ( nurse )informs patients attending physician.

Results of investigations are recorded in Investigation Form with some other routine medical data.

Timetable:

18.3.2019 - 30.6.2020: Enrolling, collection of data 1.7.2020 - 30.9.2020: Finalization od database, statistic analysis 1.10.2020 - 31.1.2021: Preparation of publications 1.2. 2021 - 31.12.2021: Result presentation

ELIGIBILITY:
Inclusion Criteria:

* central venous catheter more than 48 hours in situ
* consent of a patient

Exclusion Criteria:

* technical difficulties of ultrasound machine
* unfavorable local findings - inflammation of skin, excoriation etc.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patient hospitalized in ICU, with central venous catheter inserted for more than 48 hours
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-09-18 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of catheter related thrombosis - physician and nurse | 24hours
  Diagnostic reliability of duplex ultrasonography examination of the venous system for screening of catheter-related thrombosis performed by a general nurse

CONTACTS AND LOCATIONS:
Overall Officials: Barbora Pakostová, M.D., Principal Investigator — Krajská zdravotní a.s., Masaryk Hospital
Locations (1):
- Clinic of anaesthesiology, resuscitaion and perioperative care, Masaryk Hospital,, Ústí nad Labem, Czechia

IPD SHARING:
Plan to Share IPD: Undecided